CLINICAL TRIAL: NCT05079399
Title: Biomarker of Diabetic Retinopathy
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Ashay Bhatwadekar, PhD, RPh, Associate Professor Ophthalmology, Indiana University
Other Study IDs: 11656
Record Dates: First submitted 2021-09-11; First posted 2021-10-15 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ribonucleic acid (RNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Healthy Control
  Interventions: Other: Blood draw
- Diabetes but no retinopathy
  Interventions: Other: Blood draw
- Mild non proliferative diabetic retinopathy
  Interventions: Other: Blood draw
- Moderate non proliferative diabetic retinopathy
  Interventions: Other: Blood draw
- Severe non proliferative diabetic retinopathy
  Interventions: Other: Blood draw
- Proliferative diabetic retinopathy
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Blood samples will be collected via venipuncture

SUMMARY:
Diabetic retinopathy (DR) is a complication of diabetes in which blood vessels supplying blood to the back of the eye (retina) are dysfunctional. This can lead to an improper supply of oxygen and nutrients to the retinal tissue, or it may trigger the formation of new blood vessels in response to the oxygen/nutrient deficiency. Ultimately affecting the normal vision. There is no known marker that will provide information on the health status of retinal blood vessels. Using highly specialized cells in the blood, this study will try to discover a marker of DR.

ELIGIBILITY:
Inclusion Criteria:

* Ability to cooperate with imaging procedures.
* Health status: established type 2 diabetes
* No history of panretinal photocoagulation (PRP)
* No history of treatment with intravitreal agents for past 12 months

Exclusion Criteria:

* Previous or current malignancy
* Acute or chronic infection (HIV, hepatitis B or C, tuberculosis)
* Cerebral vascular accident or cerebral vascular procedure
* Current pregnancy
* History of organ transplantation
* Presence of a graft (to avoid any effect of the graft)
* History of previous vitrectomy
* Subjects with a history of age-related macular degeneration age-related macular degeneration (AMD), glaucoma, uveitis, and branched or central vein occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit type 2 diabetes individuals with different severities of diabetic retinopathy and non-diabetes controls.
Sampling Method: Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
mRNA and miRNA sequencing of circulating angiogenic cells isolated from study participants | Baseline and change in RNA signature in follow up visit (between 3-5 years)
Surface marker expression of inflammatory markers using flow cytometry | Baseline
miRNA expression | Baseline
Epigenetic changes in circulating angiogenic cells with different severities of diabetic retinopathy | Baseline

SECONDARY OUTCOMES:
Early Treatment Diabetic Retinopathy Study (ETDRS) clinical scoring in wide-field fundus photography | Baseline and follow up visit (between 3-5 years)
  The scoring will be between 10 (no retinopathy) and 85 (advanced proliferative diabetic retinopathy). Higher score means worst outcome
Presence or absence of neovascularization and total area of non-perfusion in fluorescein angiography (FA) | Baseline and follow up visit (between 3-5 years)
Change in vessel density in optical coherence tomography angiography (OCT-A) | Baseline and follow up visit (between 3-5 years)
Change in retinal thickness in optical coherence tomography angiography (OCT-A) | Baseline and follow up visit (between 3-5 years)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Spring Mill Clinic, Carmel, Indiana
  - Eskenazi Eye Clinic, Indianapolis, Indiana
  - Glick Eye Institute, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No